CLINICAL TRIAL: NCT02582775
Title: MT2015-20: Biochemical Correction of Severe Epidermolysis Bullosa by Allogeneic Cell Transplantation and Serial Donor Mesenchymal Cell Infusions
Brief Title: MT2015-20: Biochemical Correction of Severe EB by Allo HSCT and Serial Donor MSCs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS076
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — thymoglobulin; Antilymphocyte Serum; Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- RDEB: HCT plus MSC Arm B (Experimental): Recessive dominant epidermolysis bullosa (RDEB) patients treated per study regimen on a post-transplant cyclophosphamide allogeneic hematopoietic cell transplant (HCT) platform conditioned with reduced intensity chemotherapy and low dose total body irradiation (300 cGy), followed post-HCT by serial infusions of donor-derived mesenchymal stromal cells (MSC).
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- JEB: HCT plus MSC Arm B (Experimental): Junctional epidermolysis bullosa (JEB) patient treated per study regimen on a post-transplant cyclophosphamide allogeneic hematopoietic cell transplant (HCT) platform conditioned with reduced intensity chemotherapy and low dose total body irradiation (300 cGy), followed post-HCT by serial infusions of donor-derived mesenchymal stromal cells (MSC).
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- RDEB: HCT Plus MSC Arm E (Experimental): Recessive dominant epidermolysis bullosa (RDEB) patients treated per study regimen on a post-transplant cyclophosphamide allogeneic hematopoietic cell transplant (HCT) platform conditioned with reduced intensity chemotherapy and low dose total body irradiation (400 cGy), followed post-HCT by serial infusions of donor-derived mesenchymal stromal cells (MSC).
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- HCT with 300 cGy of TBI Arm A (Experimental): Epidermolysis bullosa patients treated per study regimen with chemotherapy and stem cell transplant without mesenchymal stem cell infusions.
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- Re-Transplant Arm C (Experimental): Epidermolysis bullosa patients treated regardless of original transplant arm with re-transplant using 300 cGy of TBI.
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- HCT Arm D (Experimental): HLA-matched epidermolysis bullosa patients treated with hematopoietic cell transplant alone using 200 cGY BID of TBI (400 cGy total).
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions
- HCT Alone Arm F (Experimental): HLA-mismatched epidermolysis bullosa patients treated with hematopoietic cell transplant alone using 200 cGy BID of TBI (400 cGy total) + addition of low dose busulfan for recipients of HLA-mismatched bone marrow
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions; Drug: Busulfan
- HCT plus MSC Arm G (Experimental): HLA-mismatched epidermolysis bullosa patients treated with hematopoietic cell transplant plus serial MSC infusions using 200 cGy BID of TBI (400 cGy total) + addition of low dose busulfan for recipients of HLA-mismatched bone marrow
  Interventions: Drug: Thymoglobulin; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Bone marrow infusion; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Donor mesenchymal stem cell infusions; Drug: Busulfan

INTERVENTIONS:
Drug: Thymoglobulin — 0.5 mg/kg IV over 6 hours on day -9 and 2 mg/kg IV over 4 hours on day -8 and day -7 with premeds and solumedrol through day -2
  Other Names: ATG; anti-thymocyte globulin
Drug: Cyclophosphamide — 14.5 mg/kg IV over 1 hour day -6 and -5 50 mg/kg IV over 2 hours with mesna 40 mg/kg IV day +2 and +3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m2 IV over 60 minutes days -6 through day -2
  Other Names: fludarabine phosphate; Fludara
Radiation: Total Body Irradiation — See arm description for dosing.
  Other Names: TBI
Procedure: Bone marrow infusion — Bone marrow infusion on Day 0
  Other Names: HCT
Drug: Tacrolimus — Day +5 through day +100 with goals of 5-10 ug/L (not used for HLA-identical related donors). When used in non-MSD recipients, tapered over 6-8 weeks starting at day +100.
  Other Names: Prograf
Drug: Mycophenolate Mofetil — 15 mg/kg IV q8h (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams. Day +5 through day 35
  Other Names: MMF
Biological: Donor mesenchymal stem cell infusions — Day 60, 100 and 180 (collected during donor BM harvest for graft)
Drug: Busulfan — busulfan IV over 3 hours on days -3 and -2 for HLA-mismatched BM recipients only (Arms F and G)
  Arms: HCT Alone Arm F; HCT plus MSC Arm G

SUMMARY:
This is a single-institution, phase II study to determine the event-free survival at 1 year post allogeneic transplant and serial mesenchymal stem cell (MSC) infusions from a related donor (HLA identical, mismatched or haploidentical) or matched unrelated donor for the biochemical correction of severe epidermolysis bullosa (EB).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe form of EB characterized by collagen, laminin, integrin, keratin or plakin deficiency (by immunofluorescence staining with protein specific antibodies or Western blotting and by mutation analysis).
* Adequate organ function within 4 weeks of study registration defined as:

  * Renal: glomerular filtration rate within normal range for age
  * Hepatic: Hepatic: bilirubin, AST/ALT, ALP < 5 x upper limit of normal
  * Pulmonary: adequate pulmonary function in the opinion of the enrolling investigator
  * Cardiac: left ventricular ejection fraction ≥ 45%, normal EKG or approved by Cardiology for transplant
* Sexually active participants must agree to use adequate birth control for the during the study period (from before the start of the preparative chemotherapy through 1 year post-transplant)
* Available donor per section 5: targeted MFI < 1,000 (MFI exceeding 1000 must be approved by the PI and treatment team.)
* Voluntary written consent - adult or parent (with information sheet for minors, if applicable) prior to any research related procedures or treatment

Exclusion Criteria:

* beta 3 laminin JEB mutants
* Active untreated systemic infection at time of transplantation (including active infection with Aspergillus or other mold within 30 days)
* History of HIV infection
* Evidence of squamous cell carcinoma
* Pregnant or breast feeding. Females of child-bearing potential must have a negative pregnancy test prior to study registration as the agents administered in this study are Pregnancy Category C and D.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Tolar, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center and Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Ebens CL, McGrath JA, Tamai K, Hovnanian A, Wagner JE, Riddle MJ, Keene DR, DeFor TE, Tryon R, Chen M, Woodley DT, Hook K, Tolar J. Bone marrow transplant with post-transplant cyclophosphamide for recessive dystrophic epidermolysis bullosa expands the related donor pool and permits tolerance of nonhaematopoietic cellular grafts. Br J Dermatol. 2019 Dec;181(6):1238-1246. doi: 10.1111/bjd.17858. Epub 2019 Jun 28. PMID 30843184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The JEB subject (n=1) was enrolled on Arm B, receiving the same therapy as the RDEB subjects, but pulled out and reported separately due to the very different baseline disease course.
Period: Overall Study
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B | HCT With 300 cGy of TBI Arm A | Re-Transplant Arm C | HCT Arm D | HCT Alone Arm F | HCT Plus MSC Arm G
Started | 7 | 9 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 9 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RDEB: HCT Plus MSC B: Recessive dominant epidermolysis bullosa (RDEB) patients treated per study regimen on a post-transplant cyclophosphamide allogeneic hematopoietic cell transplant (HCT) platform conditioned with reduced intensity chemotherapy and low dose total body irradiation (300 cGy), followed post-HCT by serial infusions of donor-derived mesenchymal stromal cells (MSC).
- RDEB: HCT Plus MSC E: Recessive dominant epidermolysis bullosa (RDEB) patients treated per study regimen on a post-transplant cyclophosphamide allogeneic hematopoietic cell transplant (HCT) platform conditioned with reduced intensity chemotherapy and low dose total body irradiation (400 cGy), followed post-HCT by serial infusions of donor-derived mesenchymal stromal cells (MSC).
- Total: Total of all reporting groups
Arm/Group | RDEB: HCT Plus MSC B | RDEB: HCT Plus MSC E | JEB: HCT Plus MSC Arm B | Total
Number analyzed (Participants) | 7 | 9 | 1 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 1 | 16
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 0 | 8
  Male | 4 | 4 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 1 | 1 | 7
  Unknown or Not Reported | 1 | 8 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 9 | 0 | 15
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: An event defined as death or a 50% increase in a patient's IScoreEB from baseline
Time Frame: 1 year post-transplant
Measure: Number; unit: Count of Participants
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 7 | 9 | 1
Count of Participants | 4 | 2 | 1

2. Secondary Outcome: Change of a Patient's iscorEB
Description: iscorEB surveys are a validated, standard of care tool used to assess disease status in patients with Epidermolysis Bullosa. Measure changes in quality of life (QOL) through pain, itching, and general QOL IScorEB questionnaire. Scores can range from 16 to 112. The QOLS scores are summed so that a higher score indicates higher quality of life.
Time Frame: 1 year post-transplant
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 4 | 6 | 1
units on a scale | -10 [-10 to 112] | -24 [-24 to 112] | 110 [16 to 112]

3. Secondary Outcome: Transplant-related Mortality
Description: Cumulative incidence will be used to estimate the probability of relapse treating non-relapse death as a competing risk and transplant-related mortality conversely treating relapse as a competing risk.
Time Frame: 180 days post-transplant
Measure: Number; unit: Participants
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 7 | 9 | 1
Participants | 0 | 0 | 0

4. Secondary Outcome: Average Change in Quality of Life
Description: Measured by the Lansky or Karnofsky score (10-100). Higher scores indicate a better outcome. Midpoint of change in scores used to indicate median.
Time Frame: 1 year post-transplant
Measure: Median (Inter-Quartile Range); unit: Change in score
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 3 | 5 | 1
Change in score | 10 [10 to 100] | 0 [10 to 100] | -30 [10 to 100]

5. Secondary Outcome: Average Change in Quality of Life
Description: Measured by the Lansky or Karnofsky score (10-100). The Karnofsky Performance Scale is an assessment tool intended to gauge a patient's functional status and ability to carry out activities of daily living. Higher scores indicate a better outcome. Midpoint of change in scores used to indicate median.
Time Frame: 2 years post-transplant
Population: Participant in "JEB: HCT plus MSC Arm B" deceased at 2 year post-transplant timepoint.
Measure: Median (Inter-Quartile Range); unit: Change in score
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 3 | 4 | 0
Change in score | 10 [10 to 100] | 0 [10 to 100] |

6. Secondary Outcome: Lymphoid Chimerism
Description: Median hematopoietic cells that are of donor origin per participant.
Time Frame: Day 28, 60, 100, 180, and year 1 and 2 post-transplant
Population: Participants in "RDEB: HCT plus MSC" arm unable to be analyzed due to missed visits.
Measure: Median (Full Range); unit: Percentage of donor derived cells
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 7 | 9 | 1
Percentage of donor derived cells
  Day 28 | 100 [0 to 100] | 60 [0 to 100] | NA — Participant unable to be analyzed.
  Day 60 | 99 [0 to 100] | 78 [0 to 100] | NA — Participant unable to be analyzed.
  Day 100 | 88 [0 to 100] | 94 [0 to 100] | NA — Participant unable to be analyzed.
  Day 180: number analyzed (Participants) | 5 | 8 | 1
  Day 180 | 100 [0 to 100] | 98.5 [0 to 100] | NA — Participant unable to be analyzed.
  1 year: number analyzed (Participants) | 3 | 3 | 0
  1 year | 100 [0 to 100] | 100 [0 to 100] |
  2 years: number analyzed (Participants) | 3 | 2 | 0
  2 years | 100 [0 to 100] | 100 [0 to 100] |

7. Secondary Outcome: Myeloid Chimerism
Description: Median hematopoietic cells that are of donor origin per participant.
Time Frame: Day 28, 60, 100, 180, and year 1 and 2 post-transplant
Population: Participants in "RDEB: HCT plus MSC" arm unable to be analyzed due to missed visits.
Measure: Median (Full Range); unit: Percentage of donor derived cells
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 7 | 9 | 1
Percentage of donor derived cells
  Day 28 | 76 [0 to 100] | 95 [0 to 100] | 23 [0 to 100]
  Day 60 | 32 [0 to 100] | 96 [0 to 100] | 0 [0 to 100]
  Day 100 | 46 [0 to 100] | 96 [0 to 100] | 0 [0 to 100]
  Day 180: number analyzed (Participants) | 5 | 8 | 1
  Day 180 | 100 [0 to 100] | 97.5 [0 to 100] | 0 [0 to 100]
  1 year: number analyzed (Participants) | 3 | 3 | 0
  1 year | 100 [0 to 100] | 100 [0 to 100] |
  2 years: number analyzed (Participants) | 3 | 2 | 0
  2 years | 100 [0 to 100] | 100 [0 to 100] |

8. Secondary Outcome: Average Change of a Patient's iscorEB
Description: iscorEB surveys are a validated, standard of care tool used to assess disease status in patients with Epidermolysis Bullosa. Measure percent of changes in quality of life (QOL) through pain, itching, and general QOL IScorEB questionnaire. Scores can range from 16 to 112. The QOLS scores are summed so that a higher score indicates higher quality of life.
Time Frame: 2 year post-transplant
Population: Participant in "JEB: HCT plus MSC Arm B" deceased at 2 year post-transplant timepoint.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
Number analyzed (Participants) | 2 | 4 | 0
units on a scale | 9 [6 to 112] | -2 [16 to 112] |

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | RDEB: HCT Plus MSC Arm B | RDEB: HCT Plus MSC Arm E | JEB: HCT Plus MSC Arm B
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/9 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/9 | 0/1
Other Adverse Events (participants affected / at risk) | 2/7 | 1/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RDEB: HCT Plus MSC Arm B (N=7) | RDEB: HCT Plus MSC Arm E (N=9) | JEB: HCT Plus MSC Arm B (N=1)
Other, specify - Veno-occlusive disease (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RDEB: HCT Plus MSC Arm B (N=7) | RDEB: HCT Plus MSC Arm E (N=9) | JEB: HCT Plus MSC Arm B (N=1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT02582775/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02582775/ICF_001.pdf